CLINICAL TRIAL: NCT04702620
Title: Measurement of Expiratory Flow Variability for the Detection of Bronchospasm in Infants Using the Ventica® Device by Revenio
Acronym: VENTICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Revenio Research (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP200338
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Healthy, Wheezing, Non Wheezing Acute Respiratory Episode
Keywords: Tidal breathing, infants, reference values
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy children without symptoms: healthy children without symptoms
  Interventions: Device: Ventica® device from Revenio
- sick children without wheezing: sick children without respiratory wheezing
  Interventions: Device: Ventica® device from Revenio
- sick children with respiratory wheezing
  Interventions: Device: Ventica® device from Revenio

INTERVENTIONS:
Device: Ventica® device from Revenio — Measurement of expiratory flow variability for the detection of bronchospasm in infants

SUMMARY:
Wheezing in infants and children less than 3 years of age children is a frequent feature that might be difficult to diagnose when only the caregivers reporting is available. Indeed, in this age group the usual reversible flow limitation measure during pulmonary function testing (PFT) is missing because PFT techniques require the full patient cooperation to perform respiratory tests. Infants PFTs have been developed to measure the same indexes than those measured in adults, but they are difficult to set-up and require medication- induced sleep during day time. However, when flow limitation is sufficient it can be detected during tidal breathing as measured during spirometry using pneumotachograph (PNT). In this test, the tidal breathing flow-volume (TBFV) loop is recorded and studied using different indices to assess the airflow limitation. But, there again, when addressing infants or very young children quiet breathing can only be achieved during sleep and medication- induced sleep necessary.

Impedance pneumography (IP) is a method for measuring changes in the thoracic electrical impedance through skin electrodes, which varies as a function of lung aeration i.e. breathing. This technique has mainly been applied to monitor respiratory rate in intensive care settings, but recent technical advancements in IP signal processing and electrode placement strategy have enabled IP to be used for accurate non-invasive tidal flow signal measurement. Compared to direct PNT, high agreement in flow signal and TBFV indices has been demonstrated in young children as well as in infants, even during induced bronchoconstriction. Moreover, in overnight recordings at home, IP was found feasible for quantifying nocturnal TBFV variability in young children with lower respiratory symptoms. In this study, it was shown that preschool children with high risk of asthma present with increased variation of tidal flow profile shape, and momentarily lowered chaoticity, compared to children with lower risk of asthma.

Recently a study in Tampere University Hospital (TAUH) Allergy centre (Tampere, Finland, PSHP ethical committee code R14027, ClinicalTrials.gov code NCT02164968) finished collecting overnight TBFV using impedance pneumography on 70 young children with suspected asthma. The preliminary analysis of this data shows that the effect of asthma treatment can be seen in TBFV variability, but to assess the diagnostic capacity of this new method, healthy control sample should be collected.

The technology developed by the Finnish medical device company Revenio Research Oy enables to evaluate the variability of the expiratory flow-volume curve. It is calculate as the expiration variability index (EVI) which is decreased in case of bronchoconstriction.

In order to explore very young children (less than 3 years of age) unable to participate to any awake lung function test, we set-up a study aiming to: 1) establish reference value for EVI in healthy children 2 months to 3 years old 2) test the variation of EVI in case of acute disease with or without wheezing in this age group children.

In this observational prospective multicenter study, we will include 110 asymptomatic healthy subjects to compute reference values of EVI. We will also include 35 previously healthy subjects who have developed an acute non wheezing disease such as fever, rhinitis, otitis or bronchitis to compare their EVI to the reference values. And finally, we will recruit 35 young subjects with an acute wheezing episode. All measurements will be performed at home by the parents, except for some wheezy children who could be hospitalized. It will be proposed to record 2 consecutive nights in healthy asymptomatic children in order to evaluate the night-to-night variability which has already shown to be small in older children.

In this multicentre study 120 children will be recruited by the present study in France and the remaining 60 children in another English centre using the same design and technology.

It is expected that only children with acute wheezing episode will have a significantly low EVI compare to the reference values established by this study.

DETAILED DESCRIPTION:
Decrease airway caliber induces airflow limitation which, in turn, will determine a decrease in the tidal breathing variability. While sleeping, tidal breathing variability will not be influenced by extra-respiratory muscle activity and therefore it will describe the physiological airway caliber change.

Impedance pneumography (IP) is a method for measuring changes in the thoracic electrical impedance through skin electrodes, which varies as a function of lung aeration i.e. breathing. This technique has mainly been applied to monitor respiratory rate in intensive care settings, but recent technical advancements in IP signal processing and electrode placement strategy have enabled IP to be used for accurate non-invasive tidal flow signal measurement. Compared to direct pneumotachograph, high agreement in flow signal and tidal breathing flow-volume (TBFV) indices has been demonstrated in young children as well as in infants, even during induced bronchoconstriction. Moreover, in overnight recordings at home, IP was found feasible for quantifying nocturnal TBFV variability in young children with lower respiratory symptoms. In this study, it was shown that preschool children with high risk of asthma present with increased variation of tidal flow profile.

The technology developed by the Finnish medical device company Revenio Research Oy enables to evaluate the variability of the expiratory flow-volume curve. It is calculate as the expiration variability index (EVI) which is decreased in case of bronchoconstriction, and momentarily lowered chaoticity, compared to children with lower risk of asthma.

We hypothesize that EVI measured during natural night sleep in children under 3 years of age, could be able to detect airway obstruction and measure its resolution. In this way this technology could be useful to follow children with repeated airway obstruction (wheezing). As a first step, we set-up a study to establish reference values of EVI in children less than 3 years and look at its relevance when children are sick with or without wheezing.

The main objective of the study is to determine the reference values of EVI in healthy 2 to 36 months old children during night sleep. Primary outcome is the EVI measured using all TBFV curves recorded by Ventica® CE marked medical device (Revenio Company).

Secondary objectives are: study night-to-night IVE reproducibility over 2 consecutive nights; determine the relevance of EVI in case of wheezing or non-wheezing acute episodes; identify any environmental and anthropometric determinant of EVI; study safety and easiness of the use of the device at home by the parents. Secondary outcomes are: concordance of EVI measurements recorded 2 consecutive nights in an asymptomatic healthy child; number of nights with correct recording (at least 5 hours/night) compared to number of trials of recording; difference between values measured during an acute wheezing episode or during fever or acute rhinitis, otitis, bronchitis in previously healthy children; anthropometric data and environmental exposure of asymptomatic healthy children; questionnaire in parents to evaluate the use of the device and potential side effects.

This is a multicentre transversal cohort study conducted in healthy and sick children aged 2 to 36 months. Healthy and sick boys and girls will be recruited from the nursery of participating hospitals or, for sick children only, from the paediatric ward. Two nights recording will be proposed to asymptomatic healthy children and 1 night to sick children.

Inclusion criteria are: for all children, 2 to 36-months-olds, term birth (> 37 ga), birth weight > 3 Percentile, no hospitalisation for newborn respiratory distress, family aware of the use of the medical device, family of legal guardian consent to the study. According to the group, group 1: no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, no current acute disease, group 2: no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, presence of current non-wheezing respiratory disease or fever, group 3: presence of current wheezing episode.

Exclusion criteria are: palatine tonsils hypertrophy with respiratory consequences; apnea-hypopnea sleep syndrome; any chronic disease which could impact pulmonary function; cutaneous disease which hampers the correct positioning of the electrodes; patient having a pace-maker or any other implanted connected electronic device or other medical device (eg ECG…); for groups 1 an 2 the use of short acting bronchodilator in the previous 8 hours; daily anti-asthma medications.

No serious side-effects are expected. A spontaneous degressive flushing of the skin where the electrodes would have stood for the night might be observed.

To obtain statistical power with correct validity the inclusion of 180 children is necessary (110 asymptomatic healthy, 35 with non-wheezing disease, 35 of during a wheezing episode), but two third of this population will be included in this b-centre French study. The 60 remaining subjects will be recruited from a third English centre using the same protocol with same methodology and device. The number of children included between 2 and 12 months, 12 and 24 months, and 24 and 36 months of age will be similar.

In France 2 centres (Paris and Nancy) will include children during 18 months. Reference values will be computed according to E.M. Wright and P Royston (Simplified estimation of age-specific reference intervals for skewed data, Statistics in Medicine 1997, vol 16, 2785-2803) using STATA software. EVI values will be described according to most determinant factors (height, age, weight…).

This study is funded by the medical device fabricant Revenio Research Oy

ELIGIBILITY:
Inclusion Criteria:

* For all children, 2 to 36-months-olds, term birth (> 37 ga), birth weight > 3 Percentile, no hospitalisation for newborn respiratory distress, family aware of the use of the medical device, family of legal guardian consent to the study. According to the group, group 1: no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, no current acute disease, group 2: no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, no history of chronic rhinitis, bronchiolitis or asthma, no respiratory allergy, presence of current non-wheezing respiratory disease or fever, group 3: presence of current wheezing episode

Exclusion Criteria:

* Tonsil hypertrophy with respiratory impact
* Clinical sleep apnea syndrome (snoring or apnea noted or breathing obstructed during sleep)
* Use of rapid onset bronchodilator for less than 8 hours (except for asthmatic infants included in an exacerbation)
* Anti-asthma treatment in progress (except for asthmatic infants included during an exacerbation)
* Known chronic cardio-respiratory or other pathology that may have a respiratory impact.
* Skin pathology preventing DM placement
* Patients with a pacemaker, continuous glucose monitor, or any other connected or implanted electronic or other medical device (e.g. ECG)

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Transversal study on healthy and sick Children from 2 to 36 months involving the use of non-invasive medical device
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-03-07 (Estimated); Study Completion 2024-03-07 (Estimated)

PRIMARY OUTCOMES:
Expiration variability index (EVI) recorded during night sleep using impedance pneumography in 2 to 36 months old children | 48 hours

SECONDARY OUTCOMES:
Variability of the EVI measurement in case of wheezing or not wheezing acute episodes in 2 to 36 months old children | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Armand Trousseau Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No